CLINICAL TRIAL: NCT06346964
Title: The Effect of Health Education on Chronic Disease Management in the Elderly
Brief Title: Self-Care Management in Chronic Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There were not enough participants for the study.
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ayşegül Akca, Faculty of Health Science, Nursing Department, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-031
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-03

CONDITIONS: Disease Self Management
Keywords: elderly; self management; chronic disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): 6 weeks of health education will be provided to older adults. Once the intervention is completed, the scales will be re-administered face-to-face or online.
  Interventions: Other: Health education
- Control (No Intervention): No intervention has been made.

INTERVENTIONS:
Other: Health education — Health education prepared for chronic disease self-management aims to improve the health behaviors of older adults.
  Arms: Education

SUMMARY:
Self-management of chronic diseases includes treatment and adoption of healthy behaviors. The research was planned to determine the effect of health education on disease management in the elderly with chronic diseases. The research will be conducted in a parallel group, randomized controlled manner. Older adults will receive 6 weeks of health education. After the training, the scales will be re-administered face to face or online.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 65-75 age group,
* Having a chronic disease

Exclusion Criteria:

* Having vision and hearing problems
* Being 76 or older
* Having a neuro-psychiatric disease

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Disease Self-Management Scale | baseline
  The scale, developed to evaluate self-management in chronic diseases, consists of 23 items and four subscales: Self-Stigma, Coping with Stigma, Health Care Effectiveness and Treatment Compliance. Expressions on the scale are rated between 1-5; It can be converted into a 100-point system (1=0, 2=25, 3=50 and 4=75 and 5=100) to facilitate interpretation and comparison in evaluation. A high score in the Self-Stigma subscale indicates high self-stigma, a high score in the Coping with Stigma subscale indicates a high ability to cope with stigma, a high score in Health Care Effectiveness indicates high health care effectiveness, and a high score in Treatment Compliance indicates good compliance. It was determined that the 21-item scale, adapted to Turkish in 2021, showed a four-factor structure and Cronbach alpha coefficients ranged between 0.789 and 0.876.
Chronic Disease Self-Management Scale | within first week
  The scale, developed to evaluate self-management in chronic diseases, consists of 23 items and four subscales: Self-Stigma, Coping with Stigma, Health Care Effectiveness and Treatment Compliance. Expressions on the scale are rated between 1-5; It can be converted into a 100-point system (1=0, 2=25, 3=50 and 4=75 and 5=100) to facilitate interpretation and comparison in evaluation. A high score in the Self-Stigma subscale indicates high self-stigma, a high score in the Coping with Stigma subscale indicates a high ability to cope with stigma, a high score in Health Care Effectiveness indicates high health care effectiveness, and a high score in Treatment Compliance indicates good compliance. It was determined that the 21-item scale, adapted to Turkish in 2021, showed a four-factor structure and Cronbach alpha coefficients ranged between 0.789 and 0.876.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk/Turkey, Turkey (Türkiye)